CLINICAL TRIAL: NCT05598567
Title: Evaluation of Hemodynamic Parameters and Cardiac Enzyme Levels in Patients Undergoing Total Abdominal Hysterectomy Under TCI-TIVA and Sevoflurane Based General Anesthesia
Brief Title: Hemodynamic Parameters and Cardiac Enzyme Levels in Patients Undergoing General Anesthesia
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, yavuz demiraran, Professor, Duzce University
Other Study IDs: drozlemersoy4
Record Dates: First submitted 2022-10-19; First posted 2022-10-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia,General; Cardiac Event
Keywords: anesthesia, general; target controlled infusion; inhalational anesthesia; cardiac enzymes
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TCI Group: Anesthesia induction will be provided by infusion of Propofol and Remifentanil with an infusion pump device called TCI (target controlled infusion). When the bispectral index (processed EEG) levels drop below 60, rocuronium will be administered at a dose of 0.6 mg/kg, and 3 minutes after that, endotracheal intubation will be performed. Propofol and Remifentanil infusion and TCI-TIVA will be continued in the maintenance of anesthesia.
  Basal values of CK, CK-MB, Troponin-I will be studied in the preoperative period. In the postoperative period, CK, CK-MB, Troponin-I values will be studied 2 times; immediately at the end of the operation and in the 8th hour from the end of the operation.
  Interventions: Other: target controlled infusion - total intravenous general anesthesia
- Sevoflurane Group: Anesthesia induction will be provided by administration of propofol 2 mg/kg, remifentanil 1 mcg/kg . When the processed EEG levels drop below 60, rocuronium will be administered at a dose of 0.6 mg/kg. 3 minutes after that, endotracheal intubation will be performed. Conventional balanced inhalation-intravenous anesthesia will be provided by administering remifentanil at 0.05 mcg/kg/min and sevoflurane 2% in the maintenance of anesthesia.
  Basal values of CK, CK-MB, Troponin-I will be studied in the preoperative period. In the postoperative period, CK, CK-MB, Troponin-I values will be studied 2 times; immediately at the end of the operation and in the 8th hour from the end of the operation.
  Interventions: Other: sevoflurane based balanced general anesthesia

INTERVENTIONS:
Other: target controlled infusion - total intravenous general anesthesia — Both interventions are subtypes of general anesthesia.
  Groups: TCI Group
Other: sevoflurane based balanced general anesthesia — Both interventions are subtypes of general anesthesia.
  Groups: Sevoflurane Group

SUMMARY:
The goal of this observational study is to learn about the effects of total intravenous general anesthesia with target controlled infusion and sevoflurane based balanced general anesthesia on hemodynamic parameters and cardiac enzyme levels in patients undergoing total abdominal hysterectomy.

DETAILED DESCRIPTION:
Total intravenous anesthesia (TIVA) is a common anesthesia method used today as an alternative to inhalation anesthesia. Loss of consciousness is an important component of general anesthesia, in order to give the patient safe analgesia and not to remember any adverse events related to the operation.

While the depth of anesthesia can be controlled by monitoring the minimum alveolar concentration (MAK) in the ventilator devices in the modern operating room , there was no more objective method than measuring the plasma level of drugs in intravenous anesthesia. The schemes created by the anesthetists according to plasma drug levels were used when administering total intravenous anesthesia. Target Controlled Anesthesia (TCI) devices on the other hand, are pumps that have been used more frequently recently and that can deliver the required blood concentration of a drug in bolus and infusion form according to pharmacokinetic models calculated with personal data. In TCI anesthesia, intravenous infusion of anesthetics provides a more stable drug concentration in the plasma and at the site of action compared to repeated bolus techniques. Thus, it is ensured that the results such as excessively high or excessively low administration of drugs are avoided and the drug remains in the therapeutic range.

In inhalation anesthesia, anesthetic substances are absorbed from the alveoli, pass into the bloodstream and reach the brain. Tracheal intake of the anesthetic agents used in this method is rapid and the depth of anesthesia can be controlled. However , the patient should be monitored and followed up for complications . An ideal inhalation anesthetic has a minimal effect on the cardiovascular and respiratory systems and has no toxic effects on these systems. Due to these properties, the most commonly used anesthetic drugs for inhalation anesthesia today are isoflurane and sevoflurane. In terms of its cardiopulmonary effects, Sevoflurane is reported to provide faster and deeper anesthesia than other anesthetics.

Aim: In this study, the researchers aim to compare the change of cardiac enzyme levels from baseline in patients undergoing total abdominal hysterectomy under general anesthesia with TCI anesthesia and sevoflurane based balanced anesthesia.

Method: 140 patients who meet the inclusion criteria and signed informed consent will be included. All patients will be monitored with routine anesthesia monitoring and bispectral index (BIS), all parameters will be checked and recorded in 5 minute intervals throughout the operation. 70 patients will receive TCI-TIVA and 70 patients will receive sevoflurane based balanced anesthesia. Creatin kinase (CK), Creatin kinase - myoglobin binding (CK-MB), Troponin I values will be determined 3 times; before the induction of anesthesia, after the extubation of the patient at the end of the operation and 8 hours after the end of the operation.

Statistical analysis: It is planned to use 'Independent Samples t test' or 'Mann-Whitney U test' in comparison of the groups, depending on the distribution of the data. Chi-square tests will be used to examine the relationships between categorical variables. 'Repeated Measure ANOVA' will be used in the evaluation of repeated measurements. Correlations between continuous variables will be analyzed by Pearson or Spearman correlation analysis, depending on the distribution of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who will undergo Total Abdominal Hysterectomy under general anesthesia
* Patients in risk group I, II,III according to the American Society of Anesthesiologists (ASA) classification

Exclusion Criteria:

* Patients for whom Intensive Care Unit (ICU) indication is required
* Chronic obstructive pulmonary disease,
* Personal or family history of malignant hyperthermia,
* Morbid obesity,
* Alcohol or drug addiction,
* History of liver or kidney disease,
* History of cardiac surgery,
* Coronary artery disease or heart failure,
* Significant anemia or hemoglobinopathy,
* Hypotension, hypovolemia, sepsis,
* Decompensated diabetic patients,
* Those who are allergic to propofol and halogens

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 140 patients between age 18 and 80 years who meet the inclusion criteria and sign informed consent will be included.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the cardiac enzyme levels | 3 times in 24 hours in the perioperative period
  Basal values of CK, CK-MB, Troponin-I will be studied in the preoperative period. In the postoperative period, CK, CK-MB, Troponin-I values will be studied 2 times; immediately at the end of the operation and in the 8th hour from the end of the operation.
Change from baseline in the hemodynamic parameters : Systolic and diastolic blood pressures (SAP and DAP) | SAP, DAP will be checked and recorded every 5 minutes throughout the operation time: from the beginning of anesthesia induction until the end of operation, in an estimated period of up to 6 hours.
  All patients will be monitored with routine anesthesia monitoring and bispectral index: SAP and DAP in mmHg will be checked and recorded in 5 minute intervals throughout the operation.
Change from baseline in the hemodynamic parameters : Heart rate (HR) | HR will be checked and recorded every 5 minutes throughout the operation time: from the beginning of anesthesia induction until the end of operation, in an estimated period of up to 6 hours.
  All patients will be monitored with routine anesthesia monitoring and bispectral index: Heart rate (HR) in bpm , will be checked and recorded in 5 minute intervals throughout the operation.
Change from baseline in the hemodynamic parameters : Peripheral oxygen saturation (sPO2) | sPO2 will be checked and recorded every 5 minutes throughout the operation time: from the beginning of anesthesia induction until the end of operation, in an estimated period of up to 6 hours.
  All patients will be monitored with routine anesthesia monitoring and bispectral index: Peripheral oxygen saturation (sPO2) in percent (%) will be checked and recorded in 5 minute intervals throughout the operation.
Change from baseline in the hemodynamic parameters : Bispectral index (BIS) | BIS in percent (%) will be checked and recorded every 5 minutes throughout the operation time: from the beginning of anesthesia induction until the end of operation, in an estimated period of up to 6 hours.
  All patients will be monitored with routine anesthesia monitoring and bispectral index: Bispectral index (BİS) will be checked and recorded in 5 minute intervals throughout the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Demiraran, Study Chair — Düzce University Faculty of Medicine
Locations (1):
- Duzce University Faculty of Medicine, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No